CLINICAL TRIAL: NCT00831805
Title: Impact of a Geriatric Mobile Unit on the Screening of Psycho-cognitive Troubles in Internal Medicine Departments and Circumstances of Calling in This Unit.
Brief Title: Screening of Psycho-cognitive Troubles in Elderly Patients
Acronym: EMG
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: ID RCB : 2008-A01107-48
Record Dates: First submitted 2008-12-08; First posted 2009-01-29 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2008-12

CONDITIONS: Psycho-cognitive Troubles
Keywords: geriatrics; psycho-cognitive troubles; elderly; mobile unit; elderly patients

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main objective of the study is to assess the rate of patients with psycho-cognitive troubles among hospitalised elderly patients.

DETAILED DESCRIPTION:
It also aims to assess this rate among patients 1) when the geriatrics mobile unit is involved in the screening of these troubles and 2) when it is not.

All the patients (75 and older) hospitalised in the internal medicine department of a suburban Parisian hospital are included in the study and their psycho-cognitive functions assessed by a geriatrics physician, using 3 validated tests.

The result of this screening provides the rate of psycho-cognitive troubles among patients that would not have been tested by a geriatrics physician in usual care. It assesses the interest of a systematic evaluation of elderly patients by the geriatric mobile unit.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 75 years old or more
* hospitalised in internal medicine

Exclusion Criteria:

* patient confused (interference with the assessment of psycho-cognitive functions)
* diagnosis of dementia at admission
* refusal of the patient or close relative for participating in the study
* poor understanding of French language
* hospitalisation for less than 3 nights

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: elderly patients hospitalised in the internal medicine department of a suburban Parisian hopital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2008-12; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
rate of patients with psycho-cognitive troubles among hospitalised elderly patients | 1 day

SECONDARY OUTCOMES:
rates of patients with psycho-cognitive troubles 1) when the geriatrics mobile unit is involved in the screening of these troubles and 2) when it is not; and comparison of these rates | 1 day
comparison of the rates of diagnosed dementia among 300 hospitalised patients, between 2006 and 2008 (before and after the creation of the geriatric mobile unit) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Charru, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Louis Mourier, Assistance Publique Hopitaux de Paris, Colombes, France